CLINICAL TRIAL: NCT04587583
Title: WeCareAdvisor: A Web-Based Tool to Improve Quality of Life for Military Veterans With Dementia and Their Caregivers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Frederic C. Blow, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00117707; W81XWH-16-1-0551 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dementia; Caregiver; Memory Disorders; Alzheimer Disease; Behavioral Symptoms
MeSH Terms: conditions — Dementia; Memory Disorders; Alzheimer Disease; Behavioral Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WeCareAdvisor (Active Comparator): immediate use of the WeCareAdvisor tool for a 1 month period
  Interventions: Behavioral: WeCareAdvisor
- WeCareAdvisor after 1 month (Active Comparator): after a wait period of 1 month, use of the WeCareAdvisor tool for a 1 month period
  Interventions: Behavioral: WeCareAdvisor

INTERVENTIONS:
Behavioral: WeCareAdvisor — Tailored, internet-based software intended to assess, manage and track behavioral symptoms and their contributing factors and to instruct dementia caregivers in problem solving approaches (tailored strategies for in-home, medication-free behavior management) to address difficult or disruptive behaviors exhibited by the person with dementia. During the testing period participants will refer to the WeCareAdvisor when behavioral challenges occur.

SUMMARY:
This research will test the WeCareAdvisor tool for family caregivers of military veterans with dementia to help caregivers assess, manage and track behavioral symptoms and their contributing factors (e.g., pain, sleep disturbance), and that provides tailored strategies for in-home, medication-free behavior management. 60 caregiver-person with dementia dyads will be recruited (30 Treatment Group, 30 Wait-List Control Group).

ELIGIBILITY:
Inclusion Criteria:

Eligible caregivers must:

* Be the primary caregiver of a military veteran with dementia for at least 6 months and planning to remain the primary caregiver for the next 2 months
* Currently living with the person they are caring for (care recipient)
* Comfortable utilizing technology (e.g. computers, tablets, the internet)
* Have access to the internet and a computer or tablet device
* Plans to live in the area for the duration of the study

Care recipients (military veteran living with dementia) must:

* Exhibit at least one or more behavioral symptoms (any behavior at any frequency)
* Receiving psychotropic medication or cognitive enhancers will not exclude the care recipient.
* Have a clinical diagnosis of dementia (any type) per caregiver report.
* Be a military veteran.

Exclusion Criteria:

* Inability to read, speak or understand English
* Lack of regular access to a telephone, internet, technology (tablet or computer)
* Caregiver is unable to use a computer or tablet
* Person with dementia is not a military veteran

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver Stress | Baseline to 2 months
  As measured by a study specific questionnaire completed by caregivers. Stress is measured on a scale of 1 to 5 where 1 is equivalent to no stress and 5 is equivalent to extreme stress.
Change in Caregiver Confidence in Managing Problematic Behavior | Baseline to 2 months
  As measured by a study specific questionnaire completed by caregivers. Confidence in managing problematic behavior is measured on a scale of 0 to 10, where a score of 0 means not confident and 10 means extremely confident
Change in Caregiver Upset | Baseline to 2 months
  As measured by a study specific questionnaire completed by caregivers. Upset is measured on a scale of 0 to 5 where 0 is equivalent to no upset and 5 is equivalent to extreme upset (midpoint is equivalent to fairly upset).

SECONDARY OUTCOMES:
Change in Caregiver Communication | Baseline to 2 months
  Caregivers rate the frequency of using six forms of negative communication (yelling, threatening, criticizing, withdrawing from patient, using harsh tone and screaming), measured on a scale of 1 to 5 where a score of 1 is never and a score of 5 is always.

OTHER OUTCOMES:
Ease of Use of the WeCareAdvisor Tool | 1 month after using WeCareAdvisor tool
  As measured by a study specific questionnaire completed by caregivers. Ease of use of the WeCareAdvisor tool is measured on a scale of 1 to 7 where 1 is equivalent to strongly disagree and 7 is equivalent to strongly agree (midpoint is equivalent to neutral).
Usefulness/ Perceived Benefit of the WeCareAdvisor Tool | 1 month after using WeCareAdvisor tool
  As measured by a study specific questionnaire completed by caregivers. Usefulness/perceived benefit of the WeCareAdvisor tool is measured on a scale of 1 to 7 where 1 is equivalent to strongly disagree and 7 is equivalent to strongly agree (midpoint is equivalent to neutral).

CONTACTS AND LOCATIONS:
Overall Officials: Frederic C Blow, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No